CLINICAL TRIAL: NCT05315193
Title: Effects of Exercise Training on Ankle-brachial Index and Quality of Life in Coronary Artery Disease Patients After Stenting.
Brief Title: Effect of Exercise Training in Coronary Artery Disease Patients After Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/01279 Umair Ahmad
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Stent Restenosis; Coronary Artery Disease
Keywords: Ankle-Brachial Index; Coronary artery diseases; Exercise training; Quality of life; Stenting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured In-patient and Home plan (Experimental): Structured In-patient and Home plan
  Interventions: Other: Structured In-patient and Home plan
- Conventional therapy (Placebo Comparator): Conventional protocol as per guidelines
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Structured In-patient and Home plan — A patient education session and a protocol comprise of 3 days. It consists of three different levels having progressive activities. The in-patient protocol will start from the day of the procedure. Each level contains 2 to 6 tasks, performed in sets of 5-10 repetitions 3 times a day. Home plan: Walking 3 days a week starting from normal pace ((RPE: 8-9) for10 minutes and progressively increased intensity and duration over the period of 12 weeks (RPE: 13-14).
  Arms: Structured In-patient and Home plan
Other: Conventional Therapy — In-Patient: Wound care, Bed mobility:
  AROMS (10 Reps*3sets*TD), Breathing Exercise (10 Reps*3sets*TD), Mobilization (Walk as per patient tolerance) Patient Education: To keep the heart healthy Diet Avoid strenuous exercise and lifting heavy objects Avoid valsalva manure, Quit smoking Lower cholesterol levels, Maintain a healthy weight Control other conditions, such as diabetes and high blood pressure Take medications as prescribed by your doctor Get regular exercise: Walking at a normal pace as per tolerance (RPE up to 10)
  Arms: Conventional therapy

SUMMARY:
To determine the effects of exercise training on ankle-brachial index and Quality of Life in coronary artery disease patients after stenting. There is a need to develop strategies, not only to prevent restenosis but also to improve patients' functional status and perception of well-being. In particular, it is not well defined whether exercise training can reduce the restenosis rate and improve the outcome after percutaneous intervention (PCI), and its effects on the Ankle-brachial index are not yet well known.

DETAILED DESCRIPTION:
The existence of PAD in patients with Coronary artery disease (CAD) remarkably increases the risk of cardiovascular morbidity and mortality. Almost half of the patients, after an initial encouraging improvement in functional capacity and quality of life (QOL) after the PCI, deal with recurrent chest pain that requires medical attention, reduces functional capacity, and creates a status of psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* GCS = 15
* Disease chronicity: 1-3 years Elective / stenting procedure
* Single or Double vessel stunting EF: 35 above

Exclusion Criteria:

* Unwilling to participate in research
* Known cases of Uncontrolled DM or HTN
* Known cases of Cognitive/memory/neurological disorders
* Known cases of any Systemic disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Ankle-brachial index | 12 weeks
  Changes From the Baseline,6th week and 12 weeks, measured through the ratio of the systolic blood pressure (SBP) measured at the ankle to that measured at the brachial artery to detect Peripheral Artery Disease. Normal Ankle-brachial index ranges from 1.0 to 1.4.
Quality of life index cardiac version -IV | 12 weeks
  Changes From the Baseline, 6th week and 12 weeks measured through Quality of life index cardiac version -IV. It consists of 70 items. Each item used a six-point Likert rating scale. Scores calculated for overall quality of life in four domains: health and functioning (15 items), social and economic (8 items), psychological/spiritual (7 items), and family (5 items). High scores indicated a better quality of life.

SECONDARY OUTCOMES:
Dyspnea | 3-5 days
  Changes From the Baseline, measured through Rose Dyspnea Scale. The scale consists of four items, with scores ranging from 0 to 4, where 0 indicates no dyspnea with activity, and increasing scores indicate greater limitations because of dyspnea.
Rate of perceived exertion (RPE) | 12 weeks
  Changes From the Baseline,6th week and 12 weeks, measured through Borg RPE scale which measures a person's perception of their effort and exertion breathlessness, and fatigue during physical work rating between 6 and 20. The higher the number, the more intense the exercise. An RPE of 6 is often referred to as just above rest, hardly any exertion, while an RPE of 20 is a maximal effort.
Forced Expiratory Volume in 1 second (FEV1) | 12 weeks
  Changes from the Baseline,6th week and 12 weeks, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 12 weeks
  Changes From the Baseline,6th week and 12 weeks, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Peshawar Institute of cardiology, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No